CLINICAL TRIAL: NCT01744067
Title: The Effects of n-3 Polyunsaturated Fatty Acids on Renal and Cardiovascular Risk Markers in Renal Transplant Recipients: a Randomized Double Blinded Placebo Controlled Intervention Study.
Brief Title: The Effects of Omega-3 Fatty Acids in Renal Transplantation
Acronym: ORENTRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Aarhus University Hospital (Other); Pronova BioPharma (Industry); South-Eastern Norway Regional Health Authority (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Ivar Eide, MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012/1419; 2012-004992-37 (EudraCT Number); 2012033 (Other Grant/Funding Number: Norway: Regional Health Authority); 2012/1419 (Other: Norway: REK)
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Disorder Related to Renal Transplantation
Keywords: Renal transplantation; Interventional study; Glomerular filtration rate; Renal function; Proteinuria; Cardiovascular risk markers; Blood pressure; Flow mediated vasodilation; Heart rate variability; Pulse wave velocity; Lipids; Blood glucose; Bone mineral density; Body composition; Fat distribution; Body mass index; Fatty acid composition; Tacrolimus pharmacokinetics; Omega-3 fatty acids; Marine n-3 fatty acids; Fatty acids; Gas chromatography; Interstitial fibrosis; Inflammation
MeSH Terms: conditions — Proteinuria; Pulmonary Fibrosis; Inflammation | interventions — Fatty Acids, Omega-3; Omacor; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 fatty acids (Active Comparator): 2,7 g omega-3 fatty acids / day: Omacor 1 g 1 capsule by mouth 3 times a day for 44 weeks.
  Interventions: Drug: Omega-3 fatty acids
- Placebo (Placebo Comparator): Placebo: 1 capsule containing 1 g of olive oil by mouth 3 times a day for 44 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omega-3 fatty acids — 2,7 g omega-3 fatty acids / day (1 capsule 3 times a day / oral administration)
  Other Names: Omacor
  Arms: Omega-3 fatty acids
Drug: Placebo — Placebo capsules 3 times a day (oral administration)
  Other Names: Olive oil
  Arms: Placebo

SUMMARY:
Omega-3 fatty acids are provided through dietary intake of fish and seafood. Several dietary supplements containing omega-3 fatty acids are also commercially available. Some studies have described beneficial effects from omega-3 fatty acids, among them are anti-inflammatory, anti-thrombotic, anti-atherosclerotic, anti-arrhythmic, anti-hypertensive and lipid-modulating effects. Other studies have not confirmed these findings. This study will investigate the effects of omega-3 fatty acids on renal function and cardiovascular risk markers in renal transplant recipients.

DETAILED DESCRIPTION:
There have been few interventional studies regarding the clinical effect of omega-3 fatty acids in renal transplantation. The aim of this study is to investigate the effects of omega-3 fatty acids on renal function and cardiovascular risk markers in renal transplant recipients.

This study is a randomized double blinded placebo controlled interventional study of 132 Norwegian renal transplant recipients. It will investigate, on the one hand, the effect of omega-3 fatty acids on renal function and, on the other, the effect of omega-3 fatty acids on cardiovascular risk markers in renal transplant recipients.

8 weeks after transplantation, if renal function has stabilized, patients with a eGFR>30 will be randomized to receive either 2,7 g eicosapentaenoic plus docosahexaenoic acid (3 capsules of Omacor a 1 g) daily or placebo. Baseline measurements will be performed before they start taking the study medication. The same measurements will performed again1 year after transplantation and the patients stops taking the study medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who have received a kidney transplant. Patients with a functioning kidney transplant, defined as eGFR>30 ml/min. Signed informed consent.

Exclusion Criteria:

* Patients participating in clinical trials with other investigational drugs. Patients who received a deceased donor kidney from a donor >75 years. Patients with a history of an allergic reaction or significant sensitivity to the study drug or drugs similar to the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate | 44 weeks
  Iohexol clearance

SECONDARY OUTCOMES:
Proteinuria | 44 weeks
  Both ACR and FEPR
Inflammation in the renal transplant | 44 weeks
  Degree of total inflammation in renal transplant biopsies, scores by PI and rescored by two pathologists.
Fibrosis in the renal transplant | 44 weeks
  As for inflammation
Blood pressure | 44 weeks
Heart rate variability | 44 weeks
Flow mediated dilation | 44 weeks
Pulse wave velocity and augmentation index | 44 weeks
Blood glucose | 44 weeks
  HbA1c and oral glucose tolerance test
Lipids | 44 weeks
  Total, LDL and HDL cholesterol, triglycerid and ratios
Body composition | 44 weeks
  Visceral fat volume and weight, visceral to subcutaneous fat ratio.
Bone mineral density | 44 weeks
  Regular BMD in the lumbar spine, hips, femur and arms and also selected to trabecular bone.
Body mass index | 44 weeks
Vitamin D levels | 44 weeks
Fatty acid composition in plasma and renal tissue | 44 weeks
Tacrolimus pharmacokinetics | 12 weeks
  Substudy of 15 patients, where we study tacrolimus trough levels, Tmax and AUC at the end of the ORENTRA trial, after a minimum of 4 weeks wash-out and again after 4 weeks of 2.7 g omega-3 fatty acid supplementation

OTHER OUTCOMES:
Incidence of post-transplant complications | 44 weeks + 8 weeks
Adverse events | 44 weeks + 8 weeks
Adverse reactions | 44 weeks
Frequency of clinically significant safety laboratory variables | 44 weeks
  Especially INR and tacrolimus trough concentrations. Follow-up by local nephrologist plus five Telephone Controls during follow-up.
Quality of life | 44 weeks
  The participants fill out SF-36 at baseline and the 1 year post transplant control for both safety reasons and measurement of differences between the groups with regards to quality of life.
Food questionnaire | 44 weeks
  Two specially designed food questionnaires to obtain data on dietary habits in general and type and amount of fish consumed
Comorbidity, concomitant medication and life-style factor interview | 44 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ivar A Eide, MD, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Oslo University Hospital Rikshospitalet, Oslo, * Other
  - Oslo University Hospital, Rikshospitalet, Oslo, Oslo County

REFERENCES:
- [Derived] Chan J, Eide IA, Tannaes TM, Waldum-Grevbo B, Jenssen T, Svensson M. Marine n-3 Polyunsaturated Fatty Acids and Cellular Senescence Markers in Incident Kidney Transplant Recipients: The Omega-3 Fatty Acids in Renal Transplantation (ORENTRA) Randomized Clinical Trial. Kidney Med. 2021 Oct 4;3(6):1041-1049. doi: 10.1016/j.xkme.2021.07.010. eCollection 2021 Nov-Dec. PMID 34939013
- [Derived] Eide IA, Reinholt FP, Jenssen T, Hartmann A, Schmidt EB, Asberg A, Bergan S, Brabrand K, Svensson M. Effects of marine n-3 fatty acid supplementation in renal transplantation: A randomized controlled trial. Am J Transplant. 2019 Mar;19(3):790-800. doi: 10.1111/ajt.15080. Epub 2018 Sep 22. PMID 30125457